CLINICAL TRIAL: NCT01610869
Title: Phase II, Randomised, Placebo Controlled, Multicentre, Feasibility Study of Low Dose (Metronomic) Cyclophosphamide With and Without Nintedanib (BIBF 1120) in Advanced Ovarian Cancer
Brief Title: Low Dose Cyclophosphamide +/-- Nintedanib in Advanced Ovarian Cancer
Acronym: METRO-BIBF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UCL/10/0470; 2011-005814-12 (Other Grant/Funding Number: Boehringer Ingelheim Ltd)
Record Dates: First submitted 2011-11-25; First posted 2012-06-04 (Estimated); Last update posted 2019-05-29 (Actual); Status verified 2018-10

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer
Keywords: Recurrence; Ovarian Neoplasms; Ovarian Diseases; Fallopian Tube Neoplasms; Neoplasms; Carcinoma; Neoplasms by site
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Recurrence; Ovarian Diseases; Neoplasms; Carcinoma; Neoplasms by Site | interventions — nintedanib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cyclophosphamide and BIBF-1120 (Experimental): Patients will receive oral BIBF 1120 (200mg bd) and cyclophosphamide (100mg) on a daily basis until disease progression or unacceptable toxicity.
  Interventions: Drug: BIBF 1120
- Cyclophosphamide and placebo (Placebo Comparator): Patients will receive oral BIBF 1120 (200mg bd) and placebo capsules on a daily basis until disease progression or unacceptable toxicity.
  Interventions: Drug: BIBF 1120

INTERVENTIONS:
Drug: BIBF 1120 — Patients will receive either cyclophosphamide (100mg)and oral BIBF 1120 (200mg bd) or cyclophosphamide (100mg) and placebo.
  Other Names: BIBF 1120 brand name: Nintedanib.

SUMMARY:
The primary objective is to explore the efficacy and safety of an all oral combination of BIBF 1120 (an inhibitor of angiogenic signalling) and metronomic cyclophosphamide in patients with multiply-relapsed advanced ovarian cancer, who have completed a minimum of two lines of previous chemotherapy and who for any reason are not suitable for further 'standard' intravenous chemotherapy treatments.

DETAILED DESCRIPTION:
A randomised placebo controlled double blind multi-centre phase II trial: BIBF 1120 200mg bd plus 100mg daily of oral cyclophosphamide (experimental arm) or oral cyclophosphamide 100mg daily plus placebo (control arm). Patients will receive oral BIBF 1120 and cyclophosphamide or cyclophosphamide and placebo continuously until disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects, ≥18 years, histologically proven recurrent advanced epithelial ovarian, fallopian tube or primary peritoneal carcinomas
* Have either undergone a hysterectomy or bilateral oophorectomy/salpingectomy and/or have been postmenopausal for 24 consecutive months (i.e. who have not had menses at any time in the preceding 24 consecutive months without an alternative medical cause)
* Performance status 0-2
* Adequate organ function
* Life expectancy >6 weeks
* Has received 2 or more lines of chemotherapy for ovarian cancer and patient is platinum resistant or platinum intolerant or not suitable for any further standard intravenous chemotherapy
* No previous oral cyclophosphamide, nintedanib, or other tyrosine kinase inhibitors such as cediranib but patients can have received anti-VEGF therapies such as bevacizumab as they will be stratified for this
* Measurable lesions according to RECIST 1.1 criteria or serum CA125 levels for evaluation by GCIG CA125 criteria are welcomed but not a prerequisite for inclusion as response will only be assessed for those with evaluable disease
* Able to give written informed consent and to complete QoL

Exclusion Criteria

* Carcinosarcoma or malignant tumour of non-epithelial origin (e.g. germ cell tumour, sex cord-stromal tumour) of the ovary, fallopian tube or peritoneum
* Clinically relevant non-healing wound, ulcer (intestinal tract, skin) or bone fracture
* Symptoms or signs of gastrointestinal obstruction requiring parenteral nutrition or hydration or any other GI disorders or abnormalities that would interfere with drug absorption or inability to take oral medication
* Active brain metastases (i.e. symptoms deteriorating, changing condition in < 4 weeks) or leptomeningeal disease. Trial entry is allowed if the brain metastases are stable (asymptomatic or condition stable for > 4 weeks).
* Dexamethasone for brain metastases is allowed if administered as stable dose for > 4 weeks before randomisation (if < 4 weeks then the patient is not eligible)
* Clinically relevant therapy-related toxicity from previous chemotherapy and radiotherapy
* History of major thromboembolic event within the last 6 months, such as pulmonary embolism or proximal deep vein thrombosis, unless on stable therapeutic anticoagulation (>3 months if on warfarin, PT / INR needs to be monitored regularly as per table 8.1 in protocol)
* Known inherited or acquired bleeding disorder
* Significant cardiovascular diseases, including uncontrolled hypertension, clinically relevant cardiac arrhythmia, unstable angina or myocardial infarction within the past 6 months, congestive heart failure > NYHA II, severe peripheral vascular disease, significantly relevant pericardial effusion
* History of a cerebral vascular accident, transient ischemic attack or subarachnoid hemorrhage within the past 6 months
* Radiographic evidence of cavitating or necrotic tumours with invasion of adjacent major blood vessels
* Laboratory values indicating an increased risk for adverse events:

  1. calculated GFR < 45 ml/min. Sites can use any calculation method according to local practice.
  2. absolute neutrophil count (ANC) < 1.5x109/L
  3. platelets < 100 x109/L
  4. haemoglobin < 90 g/L
  5. proteinuria CTCAE 2 or greater
  6. total bilirubin > x 2 ULN
  7. ALT and/or AST > 1.5 x ULN
  8. unless liver metastases present when ALT or AST > 2.5 ULN
  9. International normalized ratio (INR) > 2 or activated partial thromboplastin time (APTT) >1.5 x ULN in the absence of therapeutic anticoagulation. INR > 4 or APTT > 2.5 x ULN in presence of therapeutic anticoagulation
* Serious infections in particular if requiring systemic antibiotic (antimicrobial, antifungal or antiviral therapy), including hepatitis B and/or C infection, HIV- infection
* Poorly controlled diabetes mellitus or patient on sulphonylurea-type hypoglycaemics (e.g. gliclazide) as main diabetic control (as contraindicated with cyclophosphamide)
* Previous breast cancer patients are permitted only if diagnosis and any chemotherapy treatment for this was > 5 years previously and there is no evidence of metastatic breast cancer at trial entry (Please contact UCL CTC / CI if patient still on hormone treatment for breast cancer).
* Other malignancy diagnosed within the past 5 years. In exception to this rule, the following malignancies may be included:

  1. non-melanoma skin cancer (if adequately treated)
  2. cervical carcinoma in situ (if adequately treated)
  3. prior or synchronous endometrial cancer (if adequately treated), provided all of the following criteria are met: G1 or G2, no LVSI and FIGO (2010) stage IA only
* Serious illness or concomitant non-oncological disease such as neurologic, psychiatric or infectious disease or a laboratory abnormality that may increase the risk associated with study participation or study drug administration and in the judgment of the investigator would make the patient inappropriate for entry into the study
* Psychological, familial, sociological or geographical factors potentially hampering compliance with the study protocol and follow-up schedule e.g. active alcohol or drug abuse
* Any contraindications for therapy with cyclophosphamide, e.g. a history of severe hypersensitivity reactions to listed excipients for cyclophosphamide treatment with other investigational drugs
* Patients should not commence trial treatment within 6 weeks of any major surgical procedure
* Participation in another clinical trial testing a drug within the past four weeks before start of therapy or concomitantly with this trial
* Chemotherapy, including immunotherapy or monoclonal antibody treatment (VEGF) within 4 weeks of starting study treatment
* Hormone treatment for ovarian cancer within 2 weeks of starting study treatment (ongoing HRT is allowable)
* Any previous tyrosine kinase inhibitor treatment that has predominantly anti-angiogenic action
* Radiotherapy within 3 months not allowed except when given for symptom control >28d previously. All patients receiving any radiotherapy will require evidence of recurrent ovarian cancer outside the irradiated field either on imaging or via rising CA125
* Hypersensitivity to nintedanib, peanut or soya, or to any of the excipients of nintedanib

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2018-01-11 (Actual); Study Completion 2018-01-11 (Actual)

PRIMARY OUTCOMES:
Overall survival | After follow-up is complete (year 3-4 of the trial)
  To be measured in days, from the date of randomisation to the date of death.

SECONDARY OUTCOMES:
Quality of life and qualitative health data | After follow-up is complete (year 3-4 of the trial)
  Health questionnaires which record qualitative health data on the patient perspective of their illness and treatment. This will be measured on a 6 weekly basis, from baseline to the end of treatment.
Adverse events for all patients | After follow-up is complete (year 3-4 of the trial)
  Adverse events will be collected for patients in both groups during treatment and the groups compared during analysis. This will be measured on a 6 weekly basis, from baseline to the end of treatment. The first 12 patients will be assessed on a 3 weekly basis, from baseline to end of treatment.
Progression free survival | After follow-up is complete (year 3-4 of the trial)
  Progression free survival will be determined by measurement of tumour size using RECIST 1.1 at progression or by a rise in CA-125 tumour marker. Measured from the date of randomisation until date of confirmed disease progression. Tumour assessment carried out on 3 monthly basis, CA-125 carried out on 6 weekly basis.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Marcia Hall, Principal Investigator — Mount Vernon Cancer Centre
Locations (16):
- United Kingdom (16):
  - Kent Oncology Centre, Maidstone, Kent
  - Beatson West of Scotland Cancer Centre, Glasgow, Scotland
  - Velindre Hospital, Cardiff, Wales
  - Royal United Hospital, Bath
  - Addenbrookes Hospital, Cambridge
  - Royal Derby Hospital, Derby
  - Royal Surrey County Hospital, Guildford
  - St James's University Hospital, Leeds
  - Clatterbridge Centre for Oncology, Liverpool
  - Mount Vernon Hospital, London
  - Royal Marsden Hospital, London
  - St Bartholomew's Hospital, London
  - University College London Hospital (UCLH), London
  - Christie Hospital, Manchester
  - Churchill Hospital, Oxford
  - Wexham Park Hospital, Slough

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961
- [Derived] Hall MR, Dehbi HM, Banerjee S, Lord R, Clamp A, Ledermann JA, Nicum S, Lilleywhite R, Bowen R, Michael A, Feeney A, Glasspool R, Hackshaw A, Rustin G. A phase II randomised, placebo-controlled trial of low dose (metronomic) cyclophosphamide and nintedanib (BIBF1120) in advanced ovarian, fallopian tube or primary peritoneal cancer. Gynecol Oncol. 2020 Dec;159(3):692-698. doi: 10.1016/j.ygyno.2020.09.048. Epub 2020 Oct 16. PMID 33077258